CLINICAL TRIAL: NCT00946673
Title: A Phase I Trial of Vorinostat Concurrent With Stereotactic Radiotherapy in Treatment of Brain Metastases From Non-Small Cell Lung Cancer
Brief Title: Phase I Vorinostat Concurrent With Stereotactic Radiosurgery (SRS) in Brain Metastases From Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Principal Investigator, Griffith R Harsh, Professor of Neurosurgery, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUN0036
Record Dates: First submitted 2009-07-23; First posted 2009-07-27 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Brain Cancer; Neoplasm Metastasis; Lung Cancer; Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Brain Neoplasms; Neoplasm Metastasis; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Vorinostat; Radiotherapy

ARMS (1):
- vorinostat & stereotactic radiosurgery (Experimental)
  Interventions: Drug: Vorinostat; Procedure: Radiation Therapy

INTERVENTIONS:
Drug: Vorinostat — Orally up to 400 mg
Procedure: Radiation Therapy — Single fraction stereotactic radiotherapy - Standard of Care

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) of vorinostat given concurrently with stereotactic radiosurgery (SRS) to treat non-small cell lung cancer (NSCLCA) brain metastases in patient with 1-4 lesions.

ELIGIBILITY:
Inclusion Criteria:

* All patients age 18 years and older with histologically proven non-small cell lung cancer and 1-4 brain metastases, each measuring less than 2 cm will be eligible. Prior surgery or radiation is allowed as long as the target metastatic lesion(s) has not been treated with previous radiation.
* Adequate organ function (section 3.1.10).
* ECOG performance status 0-2.
* Life expectancy of >=12 weeks.
* Systemic chemotherapy washout period >=7 days.

Exclusion Criteria:

Patients who have previously been treated with whole brain irradiation, pediatric patients (age <18), pregnant women, and patients who are unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-06; Primary Completion 2014-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose of vorinostat with concurrent radiosurgery will be determined. | 30 days following Stereotactic Radiosurgery
During the expanded phase I portion of the study, the safety of the Maximum tolerated dose dose will be confirmed. | 30 days following Stereotactic Radiosurgery
The radiologic response, defined as local control and distant intra-cranial control rates at 3-months following radiotherapy, will be determined. | 3 months following Stereotactic Radiosurgery

SECONDARY OUTCOMES:
The short-term (< 30 days post-treatment) and long-term (> 30 days post-treatment) adverse effects will be determined. | 12 months
The 12-month survival rate from the date of Stereotactic Radiosurgery will be determined. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Griffith R. Harsh, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University School of Medicine, Stanford, California
  - Moffitt Cancer Center, Tampa, Florida